CLINICAL TRIAL: NCT02927236
Title: Neuroplasticity Following Theta-Burst Stimulation in Cocaine Use Disorder
Brief Title: Theta-Burst Stimulation as a Treatment for Reducing Cocaine Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate resources to complete study
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 999917002; 17-DA-N002 (Other: NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Cocaine Use Disorder; Cocaine Dependence
Keywords: Non-Invasive Brain Stimulation; Functional Magnetic Resonance Imaging (fMRI); intermittent theta burst stimulation (iTBS); transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot study: single arm; Expanded feasibility study: parallel arm
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pilot study: open label; Expanded feasibility study: double blind, sham controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Pilot Group (Experimental): Participants with cocaine dependence receive open label three daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions for up to 10 days.
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Expanded Feasibility Study (EFS): Cocaine - Active Group (Experimental): Participants with cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment for up to 10 days and fMRI brain scans.
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Expanded Feasibility Study (EFS): Cocaine - Sham Group (Sham Comparator): Participants with cocaine dependence receive three sham daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment for up to 10 days and fMRI brain scans.
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Expanded Feasibility Study (EFS): Healthy Control (Other): Healthy participants without cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment in one day and three sham daily iTBS sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment in one day with at least five days between the active and sham treatment.
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Theta burst stimulation is a type of TMS.To administer the iTBS treatment, a MagVenture MagPro 100 with MagOption (MagVenture Inc, Alpharetta, GA) machine equipped with a figure-8 active/sham coil will be used.

SUMMARY:
Objective: The goal of this clinical trial is to assess the tolerability of an accelerated intermittent theta burst stimulation (iTBS), a form of transcranial magnetic stimulation, intervention in participants with cocaine use disorder and then to determine if the intervention changes brain circuits related to cocaine use disorder and whether these changes relate to clinical outcomes.

The main questions it aims to answer are:

* Can individuals with cocaine use disorder tolerate accelerated iTBS (3 treatments per day for 10 days) (Pilot study)?
* Does iTBS (compared to sham iTBS) alter brain circuits related to cocaine use disorder (Expanded feasibility study)?

Researchers will compare individuals with cocaine use disorder to those without cocaine use disorder to identify differences at baseline, compare effects of the first day of iTBS treatment, and see if changes after treatment align brain circuits in those with cocaine use disorder more closely to patterns seen in those without cocaine use disorder.

Participants will:

* Undergo 10 days of iTBS treatment and two follow-up visits (1 week and 4 weeks after treatment) and complete questionnaires throughout to assess tolerability and drug use (Pilot study).
* Participants with cocaine use disorder will complete a characterization phase with questionnaires, two fMRI scans and a trial session of iTBS (sham or active) before the treatment phase (Expanded feasibility study).

DETAILED DESCRIPTION:
Background and objective: The goal of this clinical trial is to assess the tolerability of an accelerated intermittent theta burst stimulation (iTBS), a form of transcranial magnetic stimulation, intervention in participants with cocaine use disorder and then to determine if the intervention changes brain circuits related to cocaine use disorder and whether these changes relate to clinical outcomes.

The main questions it aims to answer are:

* Can individuals with cocaine use disorder tolerate accelerated iTBS (3 treatments per day for 10 days) (Pilot study)?
* Does iTBS (compared to sham iTBS) alter brain circuits related to cocaine use disorder (Expanded feasibility study)?

Researchers will compare individuals with cocaine use disorder to those without cocaine use disorder to identify differences at baseline, compare effects of the first day of iTBS treatment, and see if changes after treatment align brain circuits in those with cocaine use disorder more closely to patterns seen in those without cocaine use disorder.

Participants will:

* Undergo 10 days of iTBS treatment and two follow-up visits (1 week and 4 weeks after treatment) and complete questionnaires throughout to assess tolerability and drug use (Pilot study).
* Participants with cocaine use disorder will complete a characterization phase with questionnaires, two fMRI scans and a trial session of iTBS (sham or active) before the treatment phase (Expanded feasibility study).
* Participants with cocaine use disorder will complete a treatment phase with questionnaires, urine drug testing, two fMRI scans before and after the first day of treatment, ten days with three iTBS treatments (sham or active) each day (Expanded feasibility study).
* Participants with cocaine use disorder will complete a follow-up phase with contingency management for 11 weeks, follow-up fMRI scans 2 weeks and three months after the end of iTBS treatment and three monthly follow-up visits with urine drug testing and questionnaires after completion of the contingency management phase.
* Participants without cocaine use disorder will complete the same characterization phase as those with cocaine use disorder but will not receive a full treatment course of iTBS. Instead, they will complete the first treatment day twice, once with active and once with sham iTBS.

Study Population: Participants age 18 - 60 years of age (pilot study) and participants age 22 - 60 (Expanded Feasibility Study)

Study Design:

* Participants with cocaine dependence will receive open label iTBS in the pilot study
* Participants with cocaine dependence will receive active or sham iTBS in double blinded experiment in the Expanded Feasibility Study (EFS)
* Healthy Participants will complete the first treatment day twice and receive both active and sham iTBS treatment over two visits with at least five days between visits in a double blinded experiment

ELIGIBILITY:
* INCLUSION CRITERIA - PILOT PHASE: P1:

  1. Be able to give valid informed consent.
  2. Be 18 - 60 years of age.
  3. Right-handed.
  4. Be in good health.
  5. Absence of a specific learning disability, attention deficit hyperactivity disorder (ADHD) or cognitive impairment
  6. Participants will meet DSM-5 criteria for current moderate to severe substance (i.e., cocaine) use disorder, without a period of continuous abstinence lasting a one-month period over the last year, other than in a controlled environment.

EXCLUSION CRITERIA - PILOT PHASE: P1:

1. History of any neurological disorder that would increase seizure risk from iTBS such as stroke, brain lesions, previous neurosurgery, any history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month.
2. Current DSM-5 moderate-severe substance use disorder on a substance other than cocaine, nicotine, marijuana, or opiates (provided they are currently stable on Suboxone) or meeting withdrawal criteria for alcohol or a sedative/hypnotic/anxiolytic, or tolerance criteria in an individual using 3 or more days/week, regardless of diagnosis. Individuals will be considered stable on Suboxone if they have been on a stable dose for at least 2-weeks prior to consenting to 17-DA-N002 and have provided at least 3 urine specimens negative for illicit opioids over the same 2-week period (10 business days) with at least one test collected within two business days of the start of the period, one collected within three business days of the end of the period and one collected at least two days from either of the other two specimens. Urine results may be gathered at National Institute on Drug Abuse (NIDA) as part of screening or be provided by the Suboxone prescriber. Communication between the Suboxone provider and the MAI (or covering Staff Clinician) will be ongoing to establish continued illicit opioid abstinence between participant clearance and consent to 17-DA-N002. Individuals must be receiving their Suboxone as take-home doses from an external (i.e., non-NIDA-IRP) provider.
3. First-degree family history of any neurological disorder with a potentially hereditary basis, including migraines, epilepsy, or multiple sclerosis.
4. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes iTBS administration.
5. Noise-induced hearing loss or tinnitus.
6. Current use (any use in the past 4 weeks, daily use for more than a week within past 6 months) of any investigational drug or of any medications with psychotropic (e.g., benzodiazepines), anti or pro-convulsive action, or anti-coagulants. This will be determined at the discretion of the MAI.
7. Lifetime history of schizophrenia, bipolar disorder, mania, or hypomania.
8. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, mitral valve prolapse, or any heart condition currently under medical care.
9. Pregnant or lactating women or women with reproductive potential who engage in heterosexual sex that may lead to pregnancy and not using a medically acceptable form of contraception (such as birth control pills, condoms, or a diaphragm with spermicide).
10. Participation in any NIBS session (excluding the current protocol) less than two weeks ago. No NIBS exposure for treatment purposes in the last 6 months.

INCLUSION CRITERIA - EXPANDED FEASIBILITY PHASE (EFS):

1. Be able to give valid informed consent.
2. Agree to also participate in study 10-DA-N457, where characterization information is gathered and shared with this protocol.
3. Be 22 - 60 years of age.
4. Right-handed.
5. Be in good health.
6. Absence of a specific learning disability, ADHD or cognitive impairment
7. Cocaine dependent (CD) participants, and not healthy control (HC) participants, will meet Diagnostic and Statistical Manual (DSM)-5 criteria for current moderate to severe substance (i.e., cocaine) use disorder, without a period of continuous abstinence lasting a one-month period over the last year, other than in a controlled environment and currently seeking treatment. They will be using at least once a week in the month prior to enrollment.
8. Treatment seeking CD participants
9. MRI compatible

EXCLUSION -EFS

1. History of any neurological disorder that would increase seizure risk from iTBS such as stroke, brain lesions, previous neurosurgery, any history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month.
2. Current DSM-5 moderate-severe substance use disorder on a substance other than cocaine, nicotine, marijuana, or opiates (provided they are currently stable on a medication assisted treatment) or meeting withdrawal criteria for a sedative/hypnotic/anxiolytic, or tolerance criteria in an individual using 3 or more days/week, regardless of diagnosis. Individuals will be considered stable on a maintenance medication if they have been on a stable dose for at least 2-weeks prior to consenting to 17-DA-N002 and have provided at least 3 urine specimens negative for illicit opioids over the same 2-week period (10 business days) with at least one test collected within two business days of the start of the period, one collected within three business days of the end of the period and one collected at least two days from either of the other two specimens. Urine results may be gathered at NIDA as part of screening or be provided by the buprenorphine maintenance prescriber. Communication between the maintenance provider and the MAI (or covering Staff Clinician) will be ongoing to establish continued illicit opioid abstinence between participant clearance and consent to 17-DA-N002.
3. HC participants will not currently meet DSM-5 criteria for moderate to severe substance use disorder (excluding nicotine), and in the past, will not meet DSM-5 criteria for moderate to severe substance use disorder for cannabis or alcohol in the past 5 years or ever for other illicit substances. HC will not meet current withdrawal criteria for alcohol or sedative/hypnotics/anxiolytics, or tolerance criteria in an individual using 3 or more days/week. Urine toxicology positive for any illicit substance inconsistent with history given will also be exclusionary.
4. First-degree family history of any form of epilepsy with a potentially hereditary basis .
5. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes iTBS administration.
6. Noise-induced hearing loss or tinnitus.
7. Current use (any use in the past 4 weeks, daily use for more than a week within past 6 months) of any investigational drug or of any medications with psychotropic (e.g., benzodiazepines), anti or pro-convulsive action, or anti-coagulants. This will be determined at the discretion of the MAI.
8. Lifetime history of schizophrenia, bipolar disorder, mania, or hypomania.
9. Pregnant women or women with reproductive potential who engage in heterosexual sex that may lead to pregnancy and not using a medically acceptable form of contraception (such as birth control pills, condoms, or a diaphragm with spermicide).
10. Participation in any NIBS session less than two weeks prior to admission. No NIBS exposure for treatment purposes in the last 6 months.
11. Non-English speaking.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Yang, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steele VR, Maxwell AM, Ross TJ, Moussawi K, Abulseoud OO, Stein EA, Salmeron BJ. Report of transient events in a cocaine-dependent volunteer who received iTBS. Brain Stimul. 2018 May-Jun;11(3):631-633. doi: 10.1016/j.brs.2018.01.004. Epub 2018 Jan 31. No abstract available. PMID 29429954
- [Background] Steele VR, Rotenberg A, Philip NS, Hallett M, Stein EA, Salmeron BJ. Case report: Tremor in the placebo condition of a blinded clinical trial of intermittent theta-burst stimulation for cocaine use disorder. Front Psychiatry. 2024 Jul 9;15:1391771. doi: 10.3389/fpsyt.2024.1391771. eCollection 2024. PMID 39045554
- [Result] Steele VR, Maxwell AM, Ross TJ, Stein EA, Salmeron BJ. Accelerated Intermittent Theta-Burst Stimulation as a Treatment for Cocaine Use Disorder: A Proof-of-Concept Study. Front Neurosci. 2019 Oct 30;13:1147. doi: 10.3389/fnins.2019.01147. eCollection 2019. PMID 31736689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pilot Phase: participants complete a characterization phase prior to the treatment phase and do not proceed to the treatment phase unless they tolerate a brief trial of intermittent Theta-Burst Stimulation (iTBS) Expanded Feasibility Study (EFS) Phase: participants complete a characterization phase and do not proceed to the treatment phase unless they tolerate a brief trial of iTBS and score in the unimpaired range on Trails B, used to assess for cognitive impairment after receiving iTBS
Period: Characterization Phase
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control
Started | 19 | 4 | 3 | 19
Completed | 18 | 1 | 3 | 13
Not Completed | 1 | 3 | 0 | 6
Not completed — Physician Decision | 0 | 3 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Period: Treatment Phase
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control
Started | 14 | 1 | 2 | 12
Completed | 9 | 1 | 1 | 10
Not Completed | 5 | 0 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Follow-up Phase
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control
Started | 9 | 1 | 2 | 10
Completed | 8 | 1 | 1 | 10
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in any phase of the study.
Groups:
- Expanded Feasibility Study (EFS): Healthy Control: Healthy participants without cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double blind experiment in one day and three sham daily iTBS sessions with an inter-administration interval of at least 60-minutes between sessions in a double blind experiment in one day with at least five days between the active and sham treatment.
- Total: Total of all reporting groups
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control | Total
Number analyzed (Participants) | 19 | 4 | 3 | 19 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 4 | 3 | 19 | 45
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (8.6) | 50.25 (11.15) | 42 (8.89) | 35.7 (9.23) | 42.26 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 1 | 6 | 13
  Male | 13 | 4 | 2 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 2 | 1 | 8 | 25
  White | 3 | 2 | 2 | 6 | 13
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 4 | 3 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Cocaine Dependent Participants Who Tolerated Intermittent Theta-Burst Stimulation Sessions
Description: Number of cocaine dependent participants who tolerated the intermittent Theta-Burst Stimulation (iTBS) treatment. Participants in the pilot group had a maximum of 2 weeks and participants in the EFS group had a maximum of three weeks to complete the 10 days of treatment.
Time Frame: Up to 10 days of treatment
Population: Per protocol document, analysis applies to only participants who had cocaine dependence.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group
Number analyzed (Participants) | 14 | 1
Participants | 9 | 1

2. Primary Outcome: Change in Brain Global Efficiency After Day One of Intermittent Theta-Burst Stimulation Treatment (Acute Effect)
Description: Participants received resting brain fMRI scan followed by three iTBS sessions then a second brain fMRI scan. Analysis was done to determine if iTBS alters brain networks and calculated as the difference between global efficiency (GE) before and after the first day of iTBS (pre-post). Global efficiency is a graph-theory measure that indicates how well information can be transferred across the entire brain network. A high global efficiency indicates that information can be rapidly transmitted across different brain regions due to short average path lengths between them, suggesting a well-connected and integrated brain network. It is calculated by defining N nodes and calculating the shortest pathway between each pair of nodes. The final value is 1/N(N-1) * sum 1/shortest pathway between each pair of the N nodes. It ranges between 0 and 1 with higher values indicating greater efficiency.
Time Frame: pre/post treatment day 1.
Population: The analysis was between-subjects for cocaine dependent participants and within-subjects for healthy participants. No imaging data was collected for the Pilot arm so no results are reported.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Expanded Feasibility Study (EFS): Cocaine - Active Group: AParticipants with cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment for up to 10 days and fMRI brain scans.
- Expanded Feasibility Study (EFS): Healthy Control - Active Treatment: Healthy participants without cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in one day.
- Expanded Feasibility Study (EFS): Healthy Control - Sham Treatment: Healthy participants without cocaine dependence receive three sham daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in one day.
Arm/Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control - Active Treatment | Expanded Feasibility Study (EFS): Healthy Control - Sham Treatment
Number analyzed (Participants) | 1 | 2 | 11 | 11
unitless | -0.03716097 (0) | 0.004610517 (0.003557275) | -.01535 (0.032982662) | -0.008708172 (0.021423157)

3. Primary Outcome: Change in Brain Global Efficiency After Intermittent Theta-Burst Stimulation Treatment (iTBS) Course (Chronic Effect)
Description: Participants received baseline resting brain fMRI scan on day one and had a repeat brain fMRI two weeks after iTBS treatment course. Analysis was done to determine change in brain network with chronic treatment in cocaine dependent participants and calculated as the difference between global efficiency (GE) from baseline to post treatment (2 weeks after end of treatment). Global efficiency is a graph-theory measure that indicates how well information can be transferred across the entire brain network. A high global efficiency indicates that information can be rapidly transmitted across different brain regions due to short average path lengths between them, suggesting a well-connected and integrated brain network. It is calculated by defining N nodes and calculating the shortest pathway between each pair of nodes. The final value is 1/N(N-1) * sum 1/shortest pathway between each pair of the N nodes. It ranges between 0 and 1 with higher values indicating greater efficiency.
Time Frame: Baseline (pre-treatment) minus two weeks post treatment
Population: Analysis included only cocaine dependent participants in the Expanded Feasibility Study (EFS) arms who completed the baseline and follow up fMRI brain scans. Chronic effects of iTBS were not measured in the Pilot or in EFS healthy participants.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group
Number analyzed (Participants) | 1 | 2
unitless | -0.009259302 (0) | -0.021988865 (0.009881832)

4. Primary Outcome: Brain Global Efficiency Before Intermittent Theta-Burst Stimulation Treatment (iTBS)
Description: The brain global efficiency for cocaine dependent participants and healthy control participants at baseline (pre-treatment), prior to intermittent Theta-Burst Stimulation Treatment (iTBS). Global efficiency is a graph-theory measure that indicates how well information can be transferred across the entire brain network. A high global efficiency indicates that information can be rapidly transmitted across different brain regions due to short average path lengths between them, suggesting a well-connected and integrated brain network. It is calculated by defining N nodes and calculating the shortest pathway between each pair of nodes. The final value is 1/N(N-1) * sum 1/shortest pathway between each pair of the N nodes. It ranges between 0 and 1 with higher values indicating greater efficiency.
Time Frame: Baseline (pre-treatment)
Population: Analysis included all cocaine dependent participants (combined as one group as no intermittent Theta-Burst Stimulation (iTBS) sessions had been administered at this timepoint) and healthy control participants who had a baseline brain fMRI scan. No baseline scan was done on Pilot participants.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Expanded Feasibility Study (EFS): Cocaine Dependent Participants: Participants with cocaine dependence receive fMRI brain scan prior to intermittent Theta-Burst Stimulation (iTBS) sessions.
- Expanded Feasibility Study (EFS): Healthy Control: Healthy participants without cocaine dependence receive fMRI brain scan prior to intermittent Theta-Burst Stimulation (iTBS) sessions.
Arm/Group | Expanded Feasibility Study (EFS): Cocaine Dependent Participants | Expanded Feasibility Study (EFS): Healthy Control
Number analyzed (Participants) | 6 | 15
unitless | 0.370168044 (0.070814395) | 0.328063781 (0.035358035)

ADVERSE EVENTS:
Time Frame: Participants in the pilot phase were followed for 6 weeks. Cocaine dependent participants in the Expanded Feasibility Study (EFS) phase were followed for 6 months. Control participants in the EFS phase were participated for about two weeks.
Groups:
- Expanded Feasibility Study (EFS): Healthy Control - Active Treatment Intervention; Expanded Feasibility Study (EFS): Healthy Control - Sham Treatment Intervention: Healthy participants without cocaine dependence receive three active daily intermittent Theta-Burst Stimulation (iTBS) sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment in one day and three sham daily iTBS sessions with an inter-administration interval of at least 60-minutes between sessions in a double-blind experiment in one day with at least five days between the active and sham treatment.
Arm/Group | Pilot Group | Expanded Feasibility Study (EFS): Cocaine - Active Group | Expanded Feasibility Study (EFS): Cocaine - Sham Group | Expanded Feasibility Study (EFS): Healthy Control - Active Treatment Intervention | Expanded Feasibility Study (EFS): Healthy Control - Sham Treatment Intervention
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/4 | 0/3 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/4 | 0/3 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 0/4 | 2/3 | 2/19 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Group (N=19) | Expanded Feasibility Study (EFS): Cocaine - Active Group (N=4) | Expanded Feasibility Study (EFS): Cocaine - Sham Group (N=3) | Expanded Feasibility Study (EFS): Healthy Control - Active Treatment Intervention (N=19) | Expanded Feasibility Study (EFS): Healthy Control - Sham Treatment Intervention (N=19)
headache (Nervous system disorders) | 7 (13) | 0 (0) | 1 (3) | 1 (2) | 2 (2)
eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Eye pain during iTBS stimulation
Nervous system- other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — participant reported nightmares related to the drug cues presented during iTBS.
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported red wine-colored urine, likely related to consumption of beets and rhubarb.
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant experienced broken cuticles on fingers of right hand related to his underlying eczema.
Nervous system- other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Muscle twitching under transcranial magnetic stimulation (TMS) coil during stimulation, as expected.
tactile hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — one participant had the sensation of muscle twitching without any twitching several hours after an iTBS session. One experienced cocaine induced tactile hallucinations for the first time during the course of treatment.
scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — scalp pain under TMS coil during stimulation, as expected.
back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hang nail bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
memory loss (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — participant reported memory difficulties during a first date with someone he'd interacted online with for months and after a few beers. Resolved after the date.
muscle aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — food poisoning
tooth and ear pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — recurrence of tooth pain and tooth pain radiating to ear and unrelated to study.
tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Right hand tremor after iTBS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT02927236/Prot_SAP_001.pdf